CLINICAL TRIAL: NCT05390736
Title: Evaluating the Cost Effectiveness of STEADI Older Adult Fall Prevention in Primary Care Settings
Brief Title: Evaluating the Cost Effectiveness of STEADI
Acronym: STEADI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Opinion Research Center (Other)
Collaborators: Emory Healthcare (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dr. David Rein, Program Area Director, National Opinion Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HHSD2002013M53955B
Record Dates: First submitted 2022-05-05; First posted 2022-05-25 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Accidental Fall
MeSH Terms: interventions — Gait; Medication Review

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- STEADI Intervention (Experimental): For those assigned to the STEADI intervention arm, the clinical research nurse conducted standardized assessments to identify a patient's risk factors for falls. The STEADI assessments included: 1) a review of comorbidities; 2) medication review; 3) review of patient's falls history; 4) assessment of feet and footwear; 5) assessment of visual acuity; and 6) assessment of gait and balance; 7) review of home safety risks; and 8) assessment of potential vitamin D deficiency. Nurses would use assessment results to make recommendations which would then be relayed to the patient through their provider at their upcoming primary care visit.
  Interventions: Behavioral: Gait and balance assessment; Behavioral: Medication review; Behavioral: Comorbidity review; Behavioral: Fall history; Behavioral: Assessment of feet/footwear; Behavioral: Assessment of visual acuity; Behavioral: Home safety risk assessment; Behavioral: Vitamin D Deficiency
- Control (No Intervention): After being enrolled in the study, the patient would receive usual care from their provider.
- Physical Therapy Assessment Only (Experimental): For those assigned to the PT assessment only arm, the clinical research nurse would only conduct gait and balance assessments and would make recommendations about need for physical therapy services, conveyed to primary care provider for referrals.
  Interventions: Behavioral: Gait and balance assessment
- Medical management assessment only (Experimental): For those assign to the medical management assessment arm, only patients' medication usage would be assessed for polypharmacy (using 5 or more medications) or use of pharmaceutical classes that increase risk for falls. Recommendations for making changes to dosing levels or reducing number of medications would be conveyed to primary care provider.
  Interventions: Behavioral: Medication review

INTERVENTIONS:
Behavioral: Gait and balance assessment — Patients are given Time Up and Go (TUG) tests, 30-second chair test, and 4-stage balance test (side-by-side, instep, tandem, and one foot).
  Arms: Physical Therapy Assessment Only; STEADI Intervention
Behavioral: Medication review — Patients' medication history in the EHR is assessed for polypharmacy (using 5 or more medications concurrently) and use of medication in the following classes: tricyclic antidepressants, antihistamines, antiemetics, antipsychotics, antispasmotics, muscle relaxants, benzodiazepines, hypnotics, and opioids. The CRN confirms prescriptions with the patient. The CRN reports the medication risk in her provider report and provides medication management educational materials to the patient. At the patient's upcoming primary care visit, providers evaluated whether the medications associated with increased fall risk could be adjusted.
  Arms: Medical management assessment only; STEADI Intervention
Behavioral: Comorbidity review — The clinical research nurse reviews the patient's EHR problem list for diagnoses of comorbidities associated with increased fall risk including: cognition problems, Parkinson's disease, cardiac issues, depression, or incontinence. Comorbidities are shared with providers in the recommendation statement.
  Arms: STEADI Intervention
Behavioral: Fall history — The CRN asks how many times the patient had fallen in the past 12 months, whether those with falls sought medical attention, and if they experienced blackouts, loss of consciousness, or a broken/fractured bone(s) resulting from a fall. Fall history information is added to the provider report to increase the salience of fall prevention information.
  Arms: STEADI Intervention
Behavioral: Assessment of feet/footwear — The CRN observes or asks about the patient's current footwear, asks about foot pain or loss of sensation, and notes a diabetes diagnosis when applicable. Patient reports of foot pain, loss of sensation or diabetes result in a CRN note to the provider to examine the patient's feet and the potential need for a referral to podiatry. The CRN also reviewed a safe footwear handout with all patients regardless of their responses and emailed it to patients with other patient information following the call.
  Other Names: Podiatry / Diabetes assessment
  Arms: STEADI Intervention
Behavioral: Assessment of visual acuity — The CRN projects a Banner eye chart on Zoom for the patient to read with their contacts or glasses from five feet away for both eyes together and each eye individually. Phone patients are asked to self-report any vision problems. If either the video screening or patient self-report indicated any vision problems, the CRN notes the result and recommendation for eye care referral for the patient's provider to review and order.
  Arms: STEADI Intervention
Behavioral: Home safety risk assessment — The CRN reviews the CDC brochure "Check for Safety: A Home Fall Prevention Checklist for Older Adults" with each patient. Check for Safety asks 17 questions about the home's floors, stairs and steps, kitchen, bathrooms, and bedrooms and suggests ideas for removing or reducing fall hazards. The CRN communicates home safety risks and a recommendation for occupational therapy to the provider for indicated patients.
  Arms: STEADI Intervention
Behavioral: Vitamin D Deficiency — The CRN asks the patient if they usually take a Vitamin D supplement with their other medications. If the patient does not take a Vitamin D supplement, the CRN recommends the provider check Vitamin D levels and consider supplementation if Vitamin D levels are less than 20 ng/mL.
  Arms: STEADI Intervention

SUMMARY:
Stopping Elderly Accidents, Deaths, and Injuries (STEADI) is an intervention to prevent falls among older adults developed by the Centers for Disease Control & Prevention (CDC). Studies piloting the intervention have shown promising results; however, more evidence is needed to show that the intervention can be implemented cost-effectively on a larger scale in a real-world integrated health system. To this end, NORC partnered with Emory University School of Medicine to evaluate the effectiveness and cost-effectiveness of the STEADI intervention.

This study aims to answer the following research questions to fill remaining knowledge gaps about STEADI:

1. Does STEADI significantly reduce falls among the target population compared to the standard of care?
2. Does partial implementation of some selected STEADI modules, also significantly reduce falls among the target population as compared to the standard of care?
3. Does the net present value of falls and resulting injuries averted by STEADI implementation exceed the net present value of the costs of STEADI implementation and the incremental costs that result from it?

Using a mixture of qualitative interview and quantitative performance measures, the study evaluates and describes this case of STEADI implementation within selected primary care clinics of Emory Healthcare. NORC partnered with Emory University School of Medicine to implement different aspects of STEADI in a real-world primary care setting, document experiences implementing the intervention, measure implementation costs, and compare the outcomes of the STEADI intervention compared to control version of the intervention.

DETAILED DESCRIPTION:
The STEADI Options Trial (STEADI Trial) is a randomized control trial implemented in five Emory Healthcare primary care clinics during September 1, 2020, and December 31, 2021. The trial compared patients who received a one-time implementation of the STEADI-based fall prevention (intervention) to a control group receiving standard care. Patients were randomized based on the provider for their next scheduled routine primary care visit. Due to the COVID-19 pandemic, investigators adapted the intervention to implement it via video or phone supported telemedicine encounters conducted by a designated project nurse.

The study contacted eligible patients, screened them for fall risk using the Stay Independent Screener, consented and enrolled patients with a fall risk, conducted intervention assessments via video or phone (with video preferred), and transferred the results of the assessments to the patient's providers for intervention at the patient's next scheduled routine primary care visits. Primary care providers outside the study team were responsible for acting on assessment information.

Investigators collected data on recruitment, assessments, health service utilization, prescriptions, fall events, implementation costs, and all-cause outpatient and inpatient charges incurred over one year using administrative and electronic health records and patient surveys.

STEADI-based fall prevention was implemented in five primary care clinics operated as part of the Emory Healthcare System selected based on the willingness of their leadership to participate, geographic and sociodemographic diversity of their patient population within the Atlanta Metro Area, and size of the geriatric population they served. The CDC was responsible for project oversight and fall prevention expertise, NORC designed the study protocol and data collection instruments and managed the project, and Emory was responsible for clinical implementation.

Emory hired three clinical research interviewers (CRIs) and a clinical research nurse (CRN) to conduct recruitment, coordination, and assessments. CRIs were responsible for screening patients for fall risk, recruiting and enrolling those at risk, scheduling STEADI assessments, and conducting pre-assessment coordination calls. The CRN was responsible for conducting assessments, providing patient education, creating recommendations based on assessment information, and disseminating those recommendations to the patient's provider. Providers were responsible for acting on recommendations through the creation of clinical referrals to services or managing medications.

Providers were randomized each week 1:1 to either intervention or control study arms based on a dice roll and then assigned patients to study arm based on their scheduled provider. Providers were re-randomized each week; however, patient assignment remained the same even if they rescheduled an appointment to another week. After randomizing, a list of patients aged 65 years and older with a non-acute clinic visit scheduled three weeks in the future along with their provider-based assignment was generated and sent to the study manager for recruitment.

Three weeks prior to their scheduled primary care visit, patients received a text message link to an online SIS, which they were requested to complete prior to their upcoming scheduled primary care visit. Patients who screened at risk via the online SIS and patients who did not complete it were contacted by the study's CRIs up to three times before their primary care visit. Once reached, CRIs administered the SIS to patients who did not complete it online to determine eligibility based on fall risk. Patients with fall risk ascertained online or by phone were asked if they had 1) a computer/tablet/or phone with a camera and internet, or if not if they could participate by phone 2) space for a clear hallway and corner in their home, and 3) someone nearby they could call upon for help during the assessment. Patients who answered yes were then asked to provide informed consent to participate in the study.

Patients in the STEADI treatment groups were called by CRIs to evaluate whether their home was safe for the assessment and provided setup instructions based on a script. During this call, CRIs confirmed the patient had a stable internet connection and was able to start the video conferencing software (Zoom), and had a 10 foot path for the Timed up and go (TUG) physical therapy assessment, picked a corner for the 4-stage balance physical therapy assessment, and had an appropriate chair and wall space to set the chair against for the Chair Stand physical therapy assessment.

The CRN conducted relevant assessments based on the patient's treatment assignment to identify a patient's risk factors for falls. The CRN also reviewed health education materials with the patient and sent these materials in an email follow-up. CRNs compiled assessment results, the educational materials presented to the patient, and their recommendations for referrals and care management into the patient's EHR and sent assessment results and recommendations to the provider using the EHR messaging center.

Providers in each participating clinic were informed about the study protocol, communications methods, and actions they could take to act on information contained in the CRN report. Provider actions included ordering patient referrals to physical therapy, eye care, podiatry, the dizziness clinic, and occupational therapy, reviewing and changing patient medications, and testing patients for vitamin D levels. Providers acted on CRN recommendations at their clinical discretion.

ELIGIBILITY:
Inclusion Criteria:

* With a non-acute outpatient visit scheduled at one of the five participating primary care clinics during the study period
* Stay Independent Screening (SIS) score of 4 or higher or an answer of "yes" to one of following three key questions in the SIS:

  1. "Have you fallen in the past year?"
  2. "Do you feel unsteady when standing or walking?"
  3. "Do you worry about falling?"
* English proficient
* Access to an able-bodied person to help with gait and balance assessments

Exclusion criteria:

* Evidence in medical record of severe cognitive deficiencies (such as advanced Alzheimer's or dementia).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 780 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2023-09-18 (Actual)

PRIMARY OUTCOMES:
Falls recorded in the Electronic Medical Record. | Within one year after patient completes STEADI assessment.
  Falls identified in Emory Electronic Health Record as determined by the presence of ICD-10 diagnosis codes (W00-W19).
Medically treated falls reported in patient surveys | Within one year after patient completes STEADI assessment
  Self-reports of falls that were treated in a medical setting (regardless of whether it was treated at a study affiliated site)
Non-medically treated falls reported in patient surveys | Within one year after patient completes STEADI assessment
  Self-reports of falls that were not treated in a medical setting,
Total cost of all medical services | Within one year after patient completes STEADI assessment
  Cumulative health care allowable charges (or payments if available from claims data) for all patient services as observed in electronic health records, the estimated costs of services rendered outside of Emory Healthcare, the per person cost of screening and assessment, and the per person cost of STEADI-based fall prevention implementation.

SECONDARY OUTCOMES:
Use of primary care medical services | Within one year after STEADI assessment
  Number of recorded visits with primary care providers
Use of physical therapy medical services | Within one year after STEADI assessment
  Number of PT visits recorded
Use of occupational therapy medical services | Within one year after STEADI assessment
  Number of OT visits recorded
Use of eye care services | Within one year after STEADI assessment
  Number of eye care visits
Use of podiatry services | Within one year after STEADI assessment
  Number of podiatry visits
Level of polypharmacy | Within one year after STEADI assessment.
  The total number of medications in use by patient
Benzodiazepine dosage | Within one year after STEADI assessment
  Recorded dosage for benzodiazepine in the electronic health record (0 = not taking the medication)
Opioid dosage | Within one year after STEADI assessment
  Recorded dosage for opioids in the electronic health record (0 = not taking the medication)
Antidepressant usage | Within one year after STEADI assessment
  Recorded usage of tricyclic antidepressants
Antipsychotics usage | Within one year after STEADI assessment
  Recorded usage of antipsychotics
Hypnotics usage | Within one year after STEADI assessment
  Recorded usage of hypnotics for insomnia
Antihistamine usage | Within one year after STEADI assessment
  Recorded usage of antihistamines

CONTACTS AND LOCATIONS:
Overall Officials: David Rein, PhD, Principal Investigator — National Opinion Research Center
Locations (1):
- Emory Healthcare, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be available to other researchers.

REFERENCES:
- [Derived] Rein DB, Hackney ME, Haddad YK, Sublett FA, Moreland B, Imhof L, Peterson C, Legha JK, Mark J, Vaughan CP, Johnson Ii TM, Bergen G; Emory STEADI Implementation team. Telemedicine-Based Risk Program to Prevent Falls Among Older Adults: Protocol for a Randomized Quality Improvement Trial. JMIR Res Protoc. 2024 Mar 26;13:e54395. doi: 10.2196/54395. PMID 38346180